CLINICAL TRIAL: NCT03949855
Title: Belimumab and Rituximab Compared to Rituximab Alone for the Treatment of Primary Membranous Nephropathy (ITN080AI)
Brief Title: Belimumab With Rituximab for Primary Membranous Nephropathy
Acronym: REBOOT
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Immune Tolerance Network (ITN) (Network); GlaxoSmithKline (Industry); PPD Development, LP (Industry); Rho Federal Systems Division, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DAIT ITN080AI; NIAID CRMS ID#:38478 (Other: DAIT NIAID)
Record Dates: First submitted 2019-05-13; First posted 2019-05-14 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Membranous Nephropathy; Nephrotic Syndrome
Keywords: Primary Membranous Nephropathy; nephrotic syndrome; Pharmacokinetics (PK) Analysis; Double-Blind (Masked), Placebo-Controlled Clinical Trial; Co-administered belimumab and rituximab
MeSH Terms: conditions — Glomerulonephritis, Membranous; Nephrotic Syndrome | interventions — belimumab; Rituximab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Part A: Low Proteinuria Group - Belimumab and Rituximab (Experimental): Open-label pharmacokinetics (PK) phase.
  Participants with low proteinuria classification will receive belimumab weekly subcutaneous injections (52 doses administered Week 0 to Week 51) and rituximab infusions at Weeks 4 and 6.
  Low proteinuria classification: The excretion of ≥4 to <8 g/day of protein by the kidneys in adults. (Normal in adults: 0.15 g/day).
  Interventions: Drug: Belimumab; Drug: Rituximab
- Part A :High Proteinuria Group - Belimumab and Rituximab (Experimental): Open-label pharmacokinetics (PK) phase.
  Participants with high proteinuria classification will receive belimumab weekly subcutaneous injections (52 doses administered Week 0 to Week 51) and rituximab infusions at Weeks 4 and 6.
  High proteinuria classification: The excretion of ≥8 g/day of protein by the kidneys in adults. (Normal in adults: 0.15 g/day).
  Interventions: Drug: Belimumab; Drug: Rituximab
- Part B: Belimumab and Rituximab (Experimental): Participants in the low proteinuria classification stratification, based upon Part A, and randomized to this arm, will receive subcutaneous belimumab 400 mg (two 200 mg injections) once weekly from weeks 0-3, and then 200 mg once weekly from weeks 4-51. Participants will receive rituximab infusions at Weeks 4 and 6.
  At week 30, participants will be assessed for a response to study treatment. Participants who meet at least two out of the following three criteria at week 30 will be considered to have an inadequate response to study treatment and receive a second course of rituximab (defined as 1000 mg IV given at weeks 34 and 36):
  * Anti-PLA2R level is ≥ 25% of baseline
  * Proteinuria is ≥ 50% of baseline
  * Serum albumin is < 2.8 g/dL
  Interventions: Drug: Belimumab; Drug: Rituximab
- Part B: Placebo and Rituximab (Placebo Comparator): Participants in the low proteinuria classification stratification, based upon Part A, and randomized to this arm, will receive subcutaneous belimumab placebo 400 mg (two 200 mg injections) once weekly from weeks 0-3, and then 200 mg once weekly from weeks 4-51. Participants will receive rituximab infusions at Weeks 4 and 6.
  At week 30, participants will be assessed for a response to study treatment. Participants who meet at least two out of the following three criteria at week 30 will be considered to have an inadequate response to study treatment and receive a second course of rituximab (defined as 1000 mg IV given at weeks 34 and 36):
  * Anti-PLA2R level is ≥ 25% of baseline
  * Proteinuria is ≥ 50% of baseline
  * Serum albumin is < 2.8 g/dL
  Interventions: Drug: Placebo for Belimumab; Drug: Rituximab

INTERVENTIONS:
Drug: Belimumab — Belimumab is a recombinant, human, IgG1λ monoclonal antibody.
  Belimumab will be provided as a 200 mg sterile, liquid product in a prefilled syringe. Each syringe contains 1.0 mL of 200 mg/mL belimumab. Each syringe will be a single use.
  Standard Weekly dose:
  Part A: 200 mg. administered subcutaneously. Part B: 400 mg (two 200 mg injections) from weeks 0-3, and then 200 mg from weeks 4-51, administered subcutaneously.
  Other Names: Benlysta®
  Arms: Part A :High Proteinuria Group - Belimumab and Rituximab; Part A: Low Proteinuria Group - Belimumab and Rituximab; Part B: Belimumab and Rituximab
Drug: Placebo for Belimumab — The placebo control will be provided as a sterile liquid product in a prefilled syringe. Each syringe will be of a single use.
  Standard weekly dose:
  Part A: 200 mg. administered subcutaneously. Part B: 400 mg (two 200 mg injections) from weeks 0-3, and then 200 mg from weeks 4-51, administered subcutaneously.
  Other Names: Belimumab placebo
  Arms: Part B: Placebo and Rituximab
Drug: Rituximab — Rituximab is a monoclonal antibody with specificity for CD20, a transmembrane protein expressed on B cells from the pre-B to memory cell development stages.
  Rituximab is supplied at a concentration of 10 mg/mL in either 100 mg/10 mL or 500 mg/50 mL single-use vials for infusion. It is a clear, colorless liquid.
  Dose: 1000 mg intravenously (IV), Week 4 and -6.
  Other Names: Rituxan®

SUMMARY:
The primary objective of this study is to evaluate the effectiveness of belimumab and intravenous rituximab co-administration at inducing a complete or partial remission (CR or PR) compared to rituximab alone in participants with primary membranous nephropathy.

Background:

Primary membranous nephropathy (MN) is among the most common causes of nephrotic syndrome in adults. MN affects individuals of all ages and races. The peak incidence of MN is in the fifth decade of life.

Primary MN is recognized to be an autoimmune disease, a disease where the body's own immune system causes damage to kidneys. This damage can cause the loss of too much protein in the urine.

Drugs used to treat MN aim to reduce the attack by one's own immune system on the kidneys by blocking inflammation and reducing the immune system's function. These drugs can have serious side effects and often do not cure the disease. There is a need for new treatments for MN that are better at improving the disease while reducing fewer treatment associated side effects.

In this study, researchers will evaluate if treatment with a combination of two different drugs, belimumab and rituximab, is effective at blocking the immune attacks on the kidney compared to rituximab alone. Rituximab works by decreasing a type of immune cell, called B cells. B cells are known to have a role in MN. Once these cells are removed, disease may become less active or even inactive. However, after stopping treatment, the body will make new B cells which may cause disease to become active again.

Belimumab works by decreasing the new B cells produced by the body and, may even change the type of new B cells subsequently produced. Belimumab is approved by the US Food and Drug Administration (FDA) to treat systemic lupus erythematosus (also referred to as lupus or SLE). Rituximab is approved by the FDA to treat some types of cancer, rheumatoid arthritis, and vasculitis. Neither rituximab nor belimumab is approved by the FDA to treat MN. Treatment with a combination of belimumab and rituximab has not been studied in individuals with MN, but has been tested in other autoimmune diseases, including lupus nephritis and Sjögren's syndrome.

DETAILED DESCRIPTION:
This trial is a two-part study (Part A and Part B) of adults with primary membranous nephropathy (MN), ages 18-75 inclusive. The study will be conducted at multiple sites in the United States and Canada.

Part A: Open-label Phase

Part A is an open-label, PK study to compare belimumab exposure between participants who have "low" proteinuria (≥ 4 to < 8 g/day) and "high" proteinuria (≥ 8 g/day) at Visit -1.

Initially Part A planned to enroll 20 individuals with primary MN: 10 individuals with low proteinuria and 10 individuals with high proteinuria. All Part A participants received 200 mg subcutaneous belimumab weekly, the initially approved dose of belimumab in SLE, for 52 doses (weeks 0-51). Trough serum belimumab levels would be obtained weekly following the first 4 doses of belimumab. All participants would receive rituximab 1000 mg IV at weeks 4 and 6, and are followed after the 52 week treatment period on no study medication until week 156.

Belimumab trough levels were to be analyzed after all 20 participants received the first 4 doses to compare the belimumab exposure between the low and high proteinuria groups. If the belimumab exposure was not comparable between the high and low proteinuria groups, the belimumab dose would be doubled to 400 mg/weekly for participants with high proteinuria in Part B. Dose determination for participants with high proteinuria in Part B would be made by an adjudication committee comprised of the Protocol Chair, NIAID Medical Monitor, ITN Clinical Trial Physician, and Rho Scientist, in consultation with the belimumab PK expert at GSK.

Due in part to the observed imbalance in enrollment between the high and low proteinuria groups, an ad hoc PK analysis was conducted. The serum belimumab trough levels of the first 12 participants (8 with high proteinuria and 4 with low proteinuria) who received the first 4 belimumab doses were analyzed to compare belimumab exposure between the low and high proteinuria groups.

The results of the PK analysis were reviewed by the adjudication committee, who determined that the results did not support doubling the dose of belimumab in individuals with high proteinuria nor did it identify a new proteinuria threshold that warranted an increased belimumab dose. The belimumab PK expert at GSK concurred. Thus, enrollment into Part A has been suspended, and all participants in Part B are to receive the same dose of belimumab. All participants currently enrolled in Part A continue to receive belimumab and rituximab as previously planned and are undergoing the safety assessments as presented in Appendix A.

All enrolled participants in Part A will be followed until week 156 and will be assessed for the same study endpoints as participants in Part B.

Part B: Randomized Phase

Part B is a prospective, randomized, phase II, double-blind, placebo-controlled, multicenter clinical trial in adults with primary MN to assess the effectiveness of belimumab and rituximab at treating primary MN. Part B is commencing after the completion of the ad hoc PK analysis, which did not support increasing the belimumab dose in participants with high proteinuria.

A total of 58 participants will be randomized into two treatment arms.

Randomization will be stratified by low (≥ 4 to < 8 g/day) and high proteinuria (≥ 8 g/day). Eleven participants who entered Part B prior to protocol version 7.0 were randomized at a 1:1 ratio; 47 participants entering at or after protocol version 7.0 will be randomized at a 3:1 ratio. A total of 41 participants are projected to be enrolled in the belimumab and rituximab arm and 17 participants in the belimumab placebo and rituximab arm. The effectiveness of belimumab with rituximab will be evaluated using a hybrid control arm that combines participants who receive belimumab placebo and rituximab in this study and the subgroup of subjects with primary MN in the MENTOR trial who were anti-PLA2R positive at baseline and received rituximab alone. The randomized arms will also be used to evaluate the safety of adding belimumab to rituximab in primary MN and to support mechanistic studies.

Participants randomized to the belimumab and rituximab arm will receive subcutaneous belimumab 400 mg (two 200 mg injections) once weekly from weeks 0-3, and then 200 mg once weekly from weeks 4-51. This dosing regimen is based on the recommended dosing of subcutaneous belimumab for lupus nephritis. Participants randomized to the belimumab placebo and rituximab arm will receive subcutaneous belimumab placebo according to the same dose and schedule.

Participants in both arms will receive rituximab 1000 mg IV at weeks 4 and 6.

At week 30, participants will be assessed for a response to study treatment. Participants who meet at least two of the following three criteria at week 30 will be considered to have an inadequate response to study treatment and, defined as fulfilling at least two of the following three criteria at week 30, will receive a second course of rituximab (defined as 1000 mg IV given at weeks 34 and 36):

* Anti-PLA2R levels is ≥ 25% of baseline
* Proteinuria is ≥ 50% of baseline
* Serum albumin is < 2.8 g/dL

After the 52 week treatment period, all participants will be followed on no study medication with assessment of the primary endpoint (CR or PR) at week 104.

The primary endpoint will be assessed at week 104 because the proteinuric response to treatment is known to lag behind the active treatment period and is recommended to be assessed at least 18 months after the initiation of therapy. There will be a tolerance endpoint at week 156 to determine if treatment with belimumab with rituximab results in a more durable remission compared to rituximab alone, and to assess the rate of relapse after having achieved complete or partial remission.

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet all of the following criteria to be eligible for this study-

1. Age 18 to 75 years inclusive
2. Diagnosis of one of the following:

   1. Primary MN confirmed by a kidney biopsy within the past 5 years
   2. Primary MN that is relapsing following a CR (Section 3.3.1) or PR (Section 3.3.2), confirmed by a kidney biopsy within the past 7 years
   3. Nephrotic syndrome with eGFR > 60 mL/min/1.73m2 and no history of immunosuppressant treatment (e.g. glucocorticoids, cyclophosphamide, cyclosporine A, tacrolimus, B-cell depleting agent) for nephrotic syndrome, and without evidence of a secondary cause of nephrotic syndrome
   4. Nephrotic syndrome and a contraindication to kidney biopsy (e.g., anticoagulation, solitary kidney, body habitus that increases the risk of biopsy, or other contraindication in the opinion of the investigator), and without evidence of a secondary cause of nephrotic syndrome
3. Serum anti-PLA2R positive
4. eGFR ≥ 30 mL/min/1.73m2 while on maximally tolerated RAS blockade
5. Proteinuria:

   1. ≥ 4 and < 8 g/day that has persisted for at least the previous 3 months while on maximally tolerated RAS blockade. Documentation of persistent proteinuria may be from a 24-hour collection or calculated from a spot urine collection. Or,
   2. ≥ 8 g/day while on maximally tolerated RAS blockade
6. Blood pressure while on maximally tolerated RAS blockade:

   1. Systolic blood pressure ≤ 140 mmHg
   2. Diastolic blood pressure ≤ 90 mmHg

Exclusion Criteria:

Subjects meeting any of the following criteria will not be eligible for this study-

1. Secondary cause of MN (e.g., SLE, drug, infection, malignancy) suggested by review of the patient's medical history and/or clinical presentation
2. Rituximab use within the previous 12 months
3. Rituximab use > 12 months ago:

   1. With an undetectable CD19 B cell count, or
   2. Did not result in a CR (Section 3.3.1) or PR (Section 3.3.2) with rituximab treatment alone (e.g., without other immunosuppressive or immunomodulatory therapy)
4. Use of anti-B cell therapy other than rituximab within the previous 12 months (or 5 half-lives, whichever is greater)
5. Cyclophosphamide use within the past 3 months
6. Use of other immunosuppressive medications such as cyclosporine or tacrolimus within the past 30 days
7. Use of systemic corticosteroids within the past 30 days
8. Use of any biologic investigational agent (defined as any drug not approved for sale in the country it is used) in the previous 12 months
9. Use of any non-biologic investigational agent in the past 30 days (or 5 half-lives, whichever is greater)
10. Poorly controlled diabetes mellitus defined as hemoglobin A1c (HbA1c) ≥ 9.0%
11. Patients with diabetic glomerulopathy on renal biopsy that is:

    1. Greater than Class I diabetic glomerulopathy, or
    2. Class I diabetic glomerulopathy with a history of poor diabetic control (e.g., HbA1c ≥ 9.0%) since time of biopsy
12. Unstable kidney function defined as > 20% decrease in eGFR during the previous 3 months due to primary MN, as determined by the site investigator in consultation with the protocol chair
13. Decrease in proteinuria by 50% or more during the previous 12 months
14. WBC count < 3.0 x 103/μl
15. Absolute neutrophil count < 1.5 x 103/μl
16. Moderately severe anemia (hemoglobin < 9 g/dL)
17. History of primary immunodeficiency
18. Serum IgA < 10 mg/dL
19. Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) ≥ 2x the upper limit of normal (ULN)
20. Positive HIV serology
21. Positive HCV serology, unless treated with anti-viral therapy with achievement of a sustained virologic response (undetectable viral load 24 weeks after cessation of therapy)
22. Evidence of current or prior infection with hepatitis B, as indicated by positive HBsAg or positive HBcAb
23. Positive QuantiFERON - TB Gold test results. PPD tuberculin test may be substituted for QuantiFERON - TB Gold test
24. History of lung disease with FVC < 70% predicted, DLCO < 70% predicted, or requiring supplemental oxygen
25. History of malignant neoplasm within the last 5 years except for basal cell or squamous cell carcinoma of the skin treated with local resection only or carcinoma in situ of the uterine cervix treated locally and with no evidence of metastatic disease for 3 years
26. Absence of individualized, age-appropriate cancer screening
27. Women of child-bearing potential who are pregnant, nursing, or unwilling to be sexually inactive or use FDA-approved contraception until week 104
28. Acute or chronic infection, including current use of suppressive therapy for chronic infection, hospitalization for treatment of infection in the past 60 days, or parenteral anti-microbial (including anti-bacterial, anti-viral, or anti-fungal agents) use in the past 60 days for infection
29. History of an anaphylactic reaction or known sensitivity or intolerance to parenteral administration of contrast agents, human or murine proteins, or monoclonal antibodies, including rituximab or belimumab
30. Evidence of serious suicide risk including any history of suicidal behavior in the last 6 months and/or any suicidal ideation in the last 2 months, or who in the investigator's judgment, poses a significant suicide risk
31. Evidence of current drug or alcohol abuse or dependence, or a history of drug or alcohol abuse or dependence in the past 12 months
32. Vaccination with a live vaccine within the past 30 days
33. Other diseases or conditions or other clinically significant abnormal laboratory value which in the opinion of the investigator would put the patient at risk or confound the results of the study
34. Inability to comply with study and follow-up procedures

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Estimated)
Dates: Start 2020-03-06 (Actual); Primary Completion 2029-03-01 (Estimated); Study Completion 2030-03-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of Participants in Complete or Partial Remission (CR or PR) at Week 104. | Week 104
  . CR is defined as proteinuria of ≤ 0.3 g/day with a serum albumin ≥ 3.5 g/dL. PR is defined as a 50% or greater decrease in proteinuria compared to baseline and proteinuria < 3.5 g/day glomerular filtration rate (eGFR) from baseline.

SECONDARY OUTCOMES:
Proportion of Participants in Complete or Partial Remission (CR or PR) at Week 52 and Week 156. | Week 52, Week 156
Proportion of Participants in Complete Remission (CR) at Week 52, Week 104 and Week 156. | Week 52, Week 104, Week 156
Proportion of Participants in PR but not CR at Week 52, Week 104, Week 156. | Week 52, Week 104, Week 156
Time to Relapse for Participants who Achieved CR or PR. | Up to 156 Weeks (3 Years)
Level of Proteinuria at Week 52, Week 104 and Week 156. | Week 52, Week 104, Week 156
Proportion of participants meeting criteria for a second course of rituximab at week 30 | Week 30
Proportion of Participants in CR or PR and Anti-PLA2R Negative at week 52, 104, and 156 | Week 52, Week 104, Week 156
Proportion of Participants in PR and Anti-PLA2R Negative at week 52, 104, and 156 | Week 52, Week 104, Week 156
Proportion of participants in PR but not CR and who are anti-PLA2R negative at week 52, 104, and 156 | Week 52, Week104, Week 156
Proportion of Participants who are Anti-PLA2R Negative at week 52, 104, and 156 | Week 52, Week104, Week 156
Quality of life at weeks 52, 104, and 156 | Week 52, Week104, Week 156
Incidence of Adverse Events (AEs). | Week 0 to Week 52
Incidence of Grade 3 or Higher Infectious Adverse Events (AEs): By Treatment Group | Week 0 to Week 52
  Reference: NCI-CTCAE manual titled, National Cancer Institute (NCI)s Common Terminology Criteria for Adverse Events Version 5.0 (published November 27, 2017).
Incidence of Arterial Thromboembolic Events: By Treatment Group | Week 0 to Week 52
  Peripheral vascular embolism, mesenteric infarct, or myocardial infarction.
Incidence of Venous Thromboembolic Events: By Treatment Group | Week 0 to Week 52
  Venous thromboembolic event (VTE) is defined as a symptomatic deep vein thrombosis (DVT): the formation of a blood clot in a deep vein, detected by systematic compression ultrasonography, symptomatic DVT, or symptomatic fatal or non-fatal pulmonary embolism (PE). An embolism is a clot in the blood that forms and blocks a blood vessel. A pulmonary embolism is a blood clot that has travelled from elsewhere in the body through the blood stream to block the main artery of the lung or one of its branches.

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Nachman, Study Chair — University of Minnesota, Department of Medicine, Division of Renal Diseases and Hypertension; Iñaki Sanz, Study Chair — Emory University, Department of Medicine, Division of Rheumatology
Locations (20):
- United States (20):
  - University of Alabama at Birmingham School of Medicine: Division of Nephrology, Birmingham, Alabama
  - University of Arkansas, Little Rock, Arkansas
  - University of California San Francisco, San Francisco, California
  - Stanford University School of Medicine: Division of Nephrology, Stanford, California
  - The Lundquist Institute for Biomedical Innovation at Harbor-UCLA Medical Center:Division of Nephrology and Hypertension, Torrance, California
  - University of Colorado, Aurora, Colorado
  - Mayo Clinic Jacksonville: Department of Nephrology and Hypertension, Jacksonville, Florida
  - University of Miami Miller School of Medicine, Div of Nephrology, Miami, Florida
  - Johns Hopkins, Baltimore, Maryland
  - National Institutes of Health Clinical Center, Bethesda, Maryland
  - University of Michigan, Ann Arbor, Michigan
  - University of Minnesota Health Clinical Research Unit, Minneapolis, Minnesota
  - Washington University in St. Louis, St Louis, Missouri
  - University of Nebraska, Omaha, Nebraska
  - Columbia University Medical Center: Division of Nephrology, New York, New York
  - University of North Carolina School of Medicine: Division of Nephrology and Hypertension, Kidney Center, Chapel Hill, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - Ohio State University Wexner Medical Center: Division of Nephrology, Columbus, Ohio
  - University of Pennsylvania: Department of Medicine: Renal-Electrolyte and Hypertension Division, Philadelphia, Pennsylvania
  - Providence Medical Research Center, Providence Health Care: Nephrology, Spokane, Washington

IPD SHARING:
Plan to Share IPD: Yes
The plan is to share data upon completion of the study in: Immunology Database and Analysis Portal (ImmPort), a long-term archive of clinical and mechanistic data from DAIT-funded grants and contracts.
Time Frame: On average, within 24 months after database lock for the trial.
Access Criteria: Open access.
URL: https://www.immport.org/home

REFERENCES:
- [Derived] Ayoub I, Nachman PH. Advances in ANCA-associated vasculitis and lupus nephritis. Nat Rev Nephrol. 2021 Feb;17(2):89-90. doi: 10.1038/s41581-020-00388-x. No abstract available. PMID 33311560
- See also: National Institute of Allergy and Infectious Diseases (NIAID) — https://www.niaid.nih.gov/
- See also: Division of Allergy, Immunology, and Transplantation (DAIT) — https://www.niaid.nih.gov/about/dait
- See also: Immune Tolerance Network (ITN) — http://www.immunetolerance.org
- See also: Visit this ITN Study website for more information — http://reboot-study.org/